CLINICAL TRIAL: NCT00424996
Title: Utility of Heidelberg Retina Tomograph in Monitoring Glaucoma Progression
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Glaucoma Research Society of Canada (Other)
Responsible Party: Principal Investigator, Graham E Trope, DR, University Health Network, Toronto
Other Study IDs: UHNToronto
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Glaucoma is a chronic disease defined by characteristic changes in the optic nerve associated initially with loss of peripheral vision and is treated by lowering intraocular (inside the eye) pressure. It has been reported that noticeable changes to the optic nerve caused by glaucoma may occur several years before changes in vision are noticed. Since changes to the optic nerve and other eye structures due to glaucoma are irreversible, it is important to develop tools for the earliest possible detection of changes due to glaucoma.

The Heidelberg Retina Tomograph (HRT) is a device that is used to produce a three-dimensional map of the optic nerve and retina, and can be used to detect changes in the optic nerve and retina over time. In previous studies, it has been shown to be useful for the detection of changes due to glaucoma. However, the HRT when compared to other techniques to evaluate the optic nerve such as stereophotography, was found to only somewhat agree.

The current study will compare HRT to stereophotography to determine how good each one is at looking and documenting changes in the optic nerve over time due to glaucoma. Using HRT to initiate early topical medication or to change management requires knowing how well HRT results predict the development of visual loss. Accordingly, the results of this study may affect the management of glaucoma patients by optimizing the follow-up of people with this condition and by initiating appropriate and more individualized treatments. Early treatment is crucial for preventing further visual loss in patients with glaucoma or ocular hypertension (high pressure inside the eye).

DETAILED DESCRIPTION:
In glaucoma, treatment decisions depend on the development of morphologic and functional damage. Therefore, damage serves as an indicator of management. Commonly, progression is determined by various perimetric techniques.

However, it has been reported that clinically detectable glaucomatous structural alteration of the ONH may precede the development of reproducible white on white and blue on yellow visual field defects by up to several years.

The HRT is a confocal scanning laser tomography device that creates a three-dimensional topographic analysis of the ONH and the peripapillary retina and includes a statistical analysis to evaluate structural change over time.

This technique showed good sensitivity and high specificity in detecting glaucoma progression when tested using computer simulation. The same good results were obtained by the same authors, in another study, in a small subgroup of 16 patients who were monitored for glaucomatous progression by both HRT and ONH stereophotographs for approximately 5.5 years.

However, in our recent retrospective study, our results demonstrated only fair agreement between HRT and clinical judgment of ONH stereophotographs for progression in glaucoma, for a mean follow-up time with HRT of 2.62 years. Although, the evaluation of the ONH stereophotographs is necessarily subjective, it is widely accepted and has been shown to be effective for evaluating change. Using the stereophotographs assessments as the "reference standard", the HRT sensitivity was 78% and the specificity to 70%. The positive predictive value of the HRT was 47.8%, while the negative predictive value was 90.3%.

According to the results of this study if the frequency of true positives and false positives does not change with longer follow-up, treatment decisions would be based on a test that may be in error 52.2% of the time.

Accordingly, our previous - and other studies - study demonstrated only fair agreement between HRT and clinical judgment of ONH stereophotographs for progression in glaucoma. At present, the available evidence does not appear to be sufficient to show that the addition of HRT improves the ability to predict the development of clinical optic disc change and/or visual field loss.

Therefore the aim of the current study is to investigate the clinical significance of the HRT in monitoring glaucoma progression. In other words we will investigate how well HRT results for glaucomatous progression are able to predict the future development of optic disc and/or visual field changes in patients with OHT and glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Best-corrected visual acuity of 20/40 or better
* Subjects determined to have OHT or glaucoma
* Spherical refraction within 6.0 D with plus or minus sphere, and cylinder within 3.0 D with plus or minus cylinder
* Subjects that show progression on the HRT
* subjects stable on ONH stereophotographs
* subjects with stable and reliable visual fields
* Subjects willing to make the required visits for the study
* Subjects tolerant to dilating drops

Exclusion Criteria:

* A suspicion or actual defect in the visual field of the eye being tested that is explained by the patient's ocular status or history, other than glaucoma
* Any history of disease or use of medication that may affect visual field reliability
* Past history of stroke or diabetic retinopathy
* Inability of the pupils to be dilated to at least 4 mm for the screening visit
* Inability to undergo either perimetry test or the ophthalmic examination
* Inability to undergo adequate or better quality stereophotographs

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University glaucoma unit
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2006-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Retinal tomography | 8 year study
  Journal of OphthalmologyVolume 2014 (2014), Article ID 987389, 12 pageshttp://dx.doi.org/10.1155/2014/987389 Clinical Significance of Optic Disc Progression by Topographic Change Analysis Maps in Glaucoma: An 8-Year Follow-Up Study D. Kourkoutas,1 Y. M. Buys,2 J. G. Flanagan,2 N. Karamaounas,1 G. Georgopoulos,3 E. Iliakis,3 M. M. Moschos,3 and G. E. Trope2

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Buys, MD, FRCSC, Principal Investigator — University of Toronto, Department of Ophthalmology; Toronto Western Hospital, Toronto, Ontario, Canada; Graham E Trope, PhD, FRCSC, Study Director — University of Toronto, Department of Ophthalmology; Toronto Western Hospital, Toronto, Ontario, Canada; John Flanagan, PhD, Study Chair — University of Toronto, Department of Ophthalmology; Toronto Western Hospital, Toronto, Ontario, Canada
Locations (1):
- University of Toronto; Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Kourkoutas D, Buys YM, Flanagan JG, Hatch WV, Balian C, Trope GE. Comparison of glaucoma progression evaluated with Heidelberg retina tomograph II versus optic nerve head stereophotographs. Can J Ophthalmol. 2007 Feb;42(1):82-8. PMID 17361246